CLINICAL TRIAL: NCT02836483
Title: A Prospective, Randomized, Open, Active-controlled, Interventional, Exploratory, Phase II Trial to Evaluate the EBA, Safety and PK of Orally Administered LCB01-0371 in Adult Patients With Smear-positive Pulmonary Tuberculosis
Brief Title: A Phase II Clinical Study of LCB01-0371 to Evaluate the EBA, Safety and PK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCB01-0371-15-2-01
Record Dates: First submitted 2016-07-05; First posted 2016-07-19 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — delpazolid; BID protein, human; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): LCB01-0371 800mg, QD
  Interventions: Drug: LCB01-0371 800mg, QD
- Group 2 (Experimental): LCB01-0371 400mg, BID
  Interventions: Drug: LCB01-0371 400mg, BID
- Group 3 (Experimental): LCB01-0371 800mg, BID
  Interventions: Drug: LCB01-0371 800mg, BID
- Group 4 (Active Comparator): Tubes 3~5Tablet, QD
  Interventions: Drug: Tubes 3~5Tablet, QD
- Group 5 (Active Comparator): Zyvox 600mg, BID
  Interventions: Drug: Zyvox 600mg, BID
- Group 6 (Experimental): LCB01-0371 1200mg, QD
  Interventions: Drug: LCB01-0371 1200mg, QD

INTERVENTIONS:
Drug: LCB01-0371 800mg, QD — Oral administration
  Other Names: LCB01-0371
  Arms: Group 1
Drug: LCB01-0371 400mg, BID — Oral administration
  Other Names: LCB01-0371
  Arms: Group 2
Drug: LCB01-0371 800mg, BID — Oral administration
  Other Names: LCB01-0371
  Arms: Group 3
Drug: Tubes 3~5Tablet, QD — Oral administration
  Other Names: Tubes Tablet
  Arms: Group 4
Drug: Zyvox 600mg, BID — Oral administration
  Other Names: Zyvox Tablet
  Arms: Group 5
Drug: LCB01-0371 1200mg, QD — Oral administration
  Other Names: LCB01-0371
  Arms: Group 6

SUMMARY:
A Prospective, Randomized, Open, Active-controlled, Interventional, Exploratory, Phase II Trial of LCB01-0371.

DETAILED DESCRIPTION:
This study is designed to explore antituberculosis of LCB01-0371 through the assess of the early bactericidal activity, safety of administration.

ELIGIBILITY:
Inclusion Criteria:

1. Korean who After listening to understand the details about the clinical trial, decided to join in the clinical study, and written consent
2. The age of consent at the time of writing, only men and women under 75 years old over 19 years old
3. The First diagnosis of tuberculosis and have not received tuberculosis treatment for TB patients

Exclusion Criteria:

1. Known history of Rifampicin or Isoniazid resistance
2. Serious TB for example tuberculous encephalomeningitis, It is impossible to participate in clinical trials
3. Known History of nontuberculous mycobacteria positive
4. Other pulmonary disease which is impossible to participate in clinical trial except TB

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
EBA0-14 | V2(Baseline, Day 1), V9(Day 15)
  The extended early bactericidal activity (extended EBA) expressed as the change of log colony forming units of sputum from baseline at Day 15

SECONDARY OUTCOMES:
EBA0-2 | V2(Baseline, Day 1), V4(Day 3)
  The standard early bactericidal activity (standard EBA) expressed as the change of log colony forming units of sputum from baseline at Day 3
EBA2-14 | V4(Day 3), V9(Day 15)
  The extended early bactericidal activity (extended EBA) expressed as the change of log colony forming units of sputum from Day 3 at Day 15
EBA2-7 | V4(Day 3), V6(Day 8)
  The extended early bactericidal activity (extended EBA) expressed as the change of log colony forming units of sputum from Day 2 at Day 8

CONTACTS AND LOCATIONS:
Overall Officials: T.S Sim, M.D., Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SM, Choi SC, Mun KR, Seo JY, Cho YL, Shim TS, Lim HS. Pharmacokinetic and Pharmacodynamic Modeling Analysis of Delpazolid (LCB01-0371) in Adult Patients with Pulmonary Tuberculosis. J Clin Pharmacol. 2024 Jul;64(7):849-859. doi: 10.1002/jcph.2424. Epub 2024 Mar 4. PMID 38436463
- [Derived] Kim JS, Kim YH, Lee SH, Kim YH, Kim JW, Kang JY, Kim SK, Kim SJ, Kang YS, Kim TH, Mok J, Byun MK, Park HJ, Joh JS, Park YB, Lim HS, Choi H, Lee SH, Kim H, Yang J, Kim H, Shen X, Alsultan A, Cho I, Geiter L, Shim TS. Early Bactericidal Activity of Delpazolid (LCB01-0371) in Patients with Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2022 Feb 15;66(2):e0168421. doi: 10.1128/AAC.01684-21. Epub 2021 Dec 6. PMID 34871098